CLINICAL TRIAL: NCT01815450
Title: BLI1100-202: BLI1100 for the Treatment of Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLI1100-202
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLI1100 (Experimental): BLI1100 topical cream
  Interventions: Drug: BLI1100
- BLI1100 - modified formulation (Experimental): BLI1100 topical cream
  Interventions: Drug: BLI1100 - modified formulation
- Placebo (Placebo Comparator): Topical cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLI1100 — BLI1100 topical cream
  Arms: BLI1100
Drug: BLI1100 - modified formulation — BLI1100 topical cream
  Arms: BLI1100 - modified formulation
Drug: Placebo — Placebo topical cream
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of BLI1100 formulations to placebo for the treatment of moderate to severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12 to 45 years of age with facial acne vulgaris
* Qualifying Investigator's Global Assessment severity score
* Qualifying number of non-inflammatory lesions
* Qualifying number of inflammatory lesions

Exclusion Criteria:

* Facial hair (beard), excessive scarring, sunburn or other disfigurement that may obscure the accurate assessment of acne grade
* Using medications that are reported to exacerbate acne
* Any clinically relevant finding at their baseline physical examination or dermatological medical history such as severe systemic diseases or diseases of the facial skin
* Have a known hypersensitivity or previous allergic reaction to any of the components
* Patients who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 369 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in total lesion count | Baseline to Week 12

SECONDARY OUTCOMES:
Percent change in total lesion count | Baseline to Week 12
Investigator's Global Assessment | 12 weeks
  Rating of overall facial acne on a 5 point scale (0=clear, 4 = severe)
Local Tolerability Score | 12 weeks
  Rating of facial symptoms on a 4 point scale (0=none, 3=severe)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (15):
- United States (15):
  - Center for Dermatology Clincal Research, Fremont, California
  - North Florida Dermatology Associates, Jacksonville, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Peachtree Dermatology Associates Research Center, Atlanta, Georgia
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Clinical Partners, Johnston, Rhode Island
  - DiscoveResearch, Bryan, Texas
  - Suzanne Bruce and Associates, Houston, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - The Education and Research Foundation, Lynchburg, Virginia
  - Women's Clinical Research Center, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington